## Project: Increasing mental health literacy and peer support among caregivers: An Electronic Painting and Peer Supportive (EPPS) Platform

Date of document: 23 April 2023

Date of upload: 6 Jan 2026



## CONSENT TO PARTICIPATE IN RESEARCH

## Increasing mental health literacy and peer support among caregivers: An Electronic Painting and Peer Supportive (EPPS) Platform

| (Ethical ap | proval reference numb | er: HSEARS 2023042 | 1001) |
|---|---|---|---|
| hereby consent to participate in the captioned research conducted by Professor Angela Leung. | | | |
| I understand that informa<br>and published. However,<br>not be revealed. | | • | |
| The procedure as set ou understand the benefit(s) a | | | • • |
| I acknowledge that I have my participation at any tire | | | re and can withdraw |
| Name of Participant | | Signature of Participant | |
| Professor Angela Name of Resea | • | Signature of | Researcher |
| Date: | | | |

Hung Hom Kowloon Hong Kong 香港九龍紅磡 Tel 電話 (852) 2766 5111 Fax 傅真 (852) 2784 3374 Email 電郵 polyu@polyu.edu.hk Website 網址 www.polyu.edu.hk